CLINICAL TRIAL: NCT02764424
Title: Pain Management in Neonatal Intensive Care Units by Studying the Autonomic Balance : Interest of the Co-evaluation of NIPE and Hetero-assessment Scale : the NIPE-DOL Study
Brief Title: Pain Management in Neonatal Intensive Care Units by Studying the Autonomic Balance
Acronym: NIPE-DOL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1600008; 1954454 (Other: CNIL)
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Premature Birth; Newborn
Keywords: Newborn; Heart Rate Variability (HRV); Analgesic Nociception Index (ANI); Autonomous Nervous System (ANS)
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm or term newborns: Preterm or term newborns, hospitalized in neonatal intensive care units of our university hospital (Saint-Etienne - France), who have to acute painful stimuli related to their care will be included in the study. This painful stress is made in the patient's usual care and is not modified by the protocol. Their stress due to the painful stimuli will be measured with different scales (2 PIPP (Premature Infant Pain Profile) and DAN (Newborn Acute Pain)) and compared with the index obtained with the NIPE (Newborn Infant Parasympathetic Evaluation - MDoloris®).
  Interventions: Device: NIPE (MDoloris®)

INTERVENTIONS:
Device: NIPE (MDoloris®) — Each file consists of a simultaneous recording of an electrocardiogram signal according to usual practice (cardiac monitor PHILIPS), coupled with a concomitant registration of NIPE (Newborn Infant Parasympathetic Evaluation - MDoloris®). The electrocardiogram signal, respiration rate, oxygen saturation (SpO2) and NIPE are recorded simultaneously on a computer with a capture card. The other indices of Heart Rate Variability will be analyzed offline.
  Other Names: Newborn Infant Parasympathetic Evaluation index

SUMMARY:
Fight against the pain caused by the disease or by the diagnostic and therapeutic procedures is a daily and essential concern for the caregiver neonatologist. The quantification of pain is needed to effectively adjust analgesic therapy and by the way, to limit side effects. Several pain scales are now validated for newborns but they are based on one-off measures and hetero assessments often dependent on many factors including the operator.

Recent developments in the real time analysis of the cardiac signal under the influence of autonomic control, have led to the development of a new painful stress index. A monitor has recently been developed by Mdoloris® company and provides an Analgesia and Nociception Index (ANI index in children and adults and NIPE index - for Newborn Infant Parasympathetic Evaluation - in newborns). It is based on the study of the heart rate variability and the variations of the sympathetic and parasympathetic indices to stimuli. The validation of this nociception index has not been validated in a neonatal unit where special attention is paid to pain control.

The main purpose of our study is to show the consistency of this NIPE index (adapted to newborns) from 2 validated pain scales routinely used in neonatology in non-sedated children, hospitalized in intensive unit and neonatal intensive care unit from the University Hospital of Saint-Etienne (France).

The study will involve 40 preterm or term newborn (i.e. with a gestational age between 26 and 42 weeks and less than 3 months of life), hospitalized in neonatal intensive care units of our university hospital (Saint-Etienne - France), who have to acute painful stimuli related to their care.

DETAILED DESCRIPTION:
Fight against the pain caused by the disease or by the diagnostic and therapeutic procedures is a daily and essential concern for the caregiver neonatologist. The quantification of pain is needed to effectively adjust analgesic therapy and by the way, to limit side effects. Several pain scales are now validated for newborns but they are based on one-off measures and hetero assessments often dependent on many factors including the operator.

Recent developments in the real time analysis of the cardiac signal under the influence of autonomic control, have led to the development of a new painful stress index. A monitor has recently been developed by Mdoloris® company and provides an Analgesia and Nociception Index (ANI index in children and adults and NIPE index - for Newborn Infant Parasympathetic Evaluation - in newborns). It is based on the study of the heart rate variability and the variations of the sympathetic and parasympathetic indices to stimuli. Clinical correlations have been completed for adult patients during or after general anesthesia. The validation of this nociception index has not been validated in a neonatal unit where special attention is paid to pain control.

The main purpose of our study is to show the consistency of this NIPE index (adapted to newborns) from 2 validated pain scales routinely used in neonatology in non-sedated children, hospitalized in intensive unit and neonatal intensive care unit from the University Hospital of Saint-Etienne (France).

The study will involve 40 preterm or term newborn (i.e. with a gestational age between 26 and 42 weeks and less than 3 months of life), hospitalized in neonatal intensive care units of our university hospital (Saint-Etienne - France), who have to acute painful stimuli related to their care.

Concurrent analysis of autonomic markers (orthosympathetic and parasympathetic indices from time or frequency domain analysis of heart rate variability) will be correlated with the NIPE index in order to study confounding factors that can induce a sympathetic stress without pain sensation and can thus change the indices of nociception.

This study based on a real-time analysis of the perception of pain for newborns is a step for the validation of this new tool that could facilitate the real-time newborn pain management. Furthermore, it will allow caregivers the opportunity to adjust therapeutics in non-communicative patients.

ELIGIBILITY:
Inclusion Criteria:

* Neonates over 26 weeks of Gestational Age, under 3 months, hospitalized in neonatal intensive care units of the university hospital of Saint-Etienne (France);
* Neonates with a potentially painful move programmed (dextro, administration of substances by intramuscular, arterial/ venipuncture, change nasogastric tube, tracheal aspirates).

Exclusion Criteria:

* Newborns sedated;
* Newborn with a treatment known to alter the sympathetic or parasympathetic activity of the autonomic nervous system.

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates over 26 weeks of Gestational Age and under 3 months hospitalized in neonatal intensive care units of the university hospital of Saint-Etienne (France) will be eligible. They will have to perform a potentially painful care (for example an administration of substances by intramuscular way) in the usual care context.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
NIPE index | Day 1
  Newborn Infant Parasympathetic Evaluation (NIPE) index obtained will be compared to the Premature Infant Pain Profile (PIPP) and ("Douleur Aiguë du Nouveau Né" - Newborn Acute Pain (DAN) scores.

SECONDARY OUTCOMES:
Orthosympathetic and parasympathetic indices | Day 1
  Compare the changes of orthosympathetic and parasympathetic indices in the time and frequency domains of heart rate variability, with respect to changes of NIPE (Newborn Infant Parasympathetic Evaluation) and PIPP-R (Premature Infant Pain Profile) / DAN (Newborn Acute Pain) scores.
Changes in the NIPE index | Day 1
  Ensure consistency of changes in levels of pain felt (PIPP score / DAN score) with changes in NIPE index, in the same patient.

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cremillieux C, Makhlouf A, Pichot V, Trombert B, Patural H. Objective assessment of induced acute pain in neonatology with the Newborn Infant Parasympathetic Evaluation index. Eur J Pain. 2018 Jul;22(6):1071-1079. doi: 10.1002/ejp.1191. Epub 2018 Mar 24. PMID 29369446